CLINICAL TRIAL: NCT00460629
Title: Specific Cellular Immunotherapy in Patients With Chronic Myeloid Leukemia After Allogeneic Stem Cell Transplantation
Brief Title: Prophylactic Transfer of Leukemia-reactive T Cells After Allogeneic Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Carl Gustav Carus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK126092000
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Adoptive immunotherapy; BCR-ABL reactive T cells; Allogeneic Transplantation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Application of activated donor T cells — Ex-vivo generated donor T cells stimulated by antigen presenting cells loaded with peptides derived from leukemia-associated antigens

SUMMARY:
Efforts to decrease the risk of GvHD by depleting T cells from the graft in CML patients have been complicated by an increased incidence of leukemia-relapse. Newer protocols using CD34+ selected hematopoietic cells from matched-sibling donors and subsequent infusion of T cells in incremental doses to treat or avoid relapse of disease seem to be more promising. In this study, we try to further optimize this approach by the prophylactic infusion of cytotoxic T cells activated ex-vivo against leukemia-associated/specific antigens using peptide-pulsed dendritic cells.

DETAILED DESCRIPTION:
The conditioning protocol contains:

Total Body Irradiation 8-12 Gy (4-6 x 2 Gy, a 2 x/die) day -9 to-7 Thiotepa 10 mg/kg (2 x 5 mg/kg) day -5 Fludarabine 200 mg/m2 (5 x 40 mg/m2) day -6 to-2 ATG Fresenius 25 mg/kg (5 x 5 mg/kg) day -6 to-2 Cyclosporine A 1 mg/kg Day -10 to-3

on day 0 CD34+ cells after immunomagnetic selection are infused. > 4 x 10e6/kg CD34 cells/kg are required.

On days 28, 56 and 112 after transplantation, cytotoxic T cells generated in-vitro are infused in patients who do not have signs of acute GvHD.

Regular follow-up compromises immune monitoring including Tetramer analyses of Peptide-reactive T cells

ELIGIBILITY:
Inclusion Criteria:

* age 18-60
* Ph+ CML
* HLA A0201, 0301, 1101, B0801
* BCR-ABL b3a2 positive
* no significant comorbidities
* resistance or intolerance of imatinib

Exclusion Criteria:

* HIV positive
* blast crisis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-03; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the infusion of in-vitro activated donor T cells | 5 years
kinetic of BCR-ABL load after transplantation | 5 years

SECONDARY OUTCOMES:
Rate of acute and chronic GvHD | 3 years
Rate of infectious complications | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bornhäuser, MD, Principal Investigator — Medical Clinic, University Hospital Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, Dresden, Germany

REFERENCES:
- [Result] Bornhauser M, Thiede C, Babatz J, Schetelig J, Illmer T, Kiani A, Platzbecker U, Herr W, Rieber EP, Ehninger G, Schmitz M. Infusion of bcr/abl peptide-reactive donor T cells to achieve molecular remission of chronic myeloid leukemia after CD34+ selected allogeneic hematopoietic cell transplantation. Leukemia. 2006 Nov;20(11):2055-7. doi: 10.1038/sj.leu.2404383. Epub 2006 Aug 31. No abstract available. PMID 16990776
- [Derived] Bornhauser M, Thiede C, Platzbecker U, Kiani A, Oelschlaegel U, Babatz J, Lehmann D, Holig K, Radke J, Tuve S, Wermke M, Wehner R, Jahnisch H, Bachmann MP, Rieber EP, Schetelig J, Ehninger G, Schmitz M. Prophylactic transfer of BCR-ABL-, PR1-, and WT1-reactive donor T cells after T cell-depleted allogeneic hematopoietic cell transplantation in patients with chronic myeloid leukemia. Blood. 2011 Jun 30;117(26):7174-84. doi: 10.1182/blood-2010-09-308569. Epub 2011 May 3. PMID 21540460